CLINICAL TRIAL: NCT00804466
Title: Epidemiologic and Molecular Features of Cervical Cancer in Nigeria - Project Itoju (Care)
Brief Title: Human Papillomavirus Epidemiology in Nigeria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 999909045; 09-C-N045
Record Dates: First submitted 2008-12-05; First posted 2008-12-08 (Estimated); Last update posted 2020-11-25 (Actual); Status verified 2019-11

CONDITIONS: Human Papillomavirus 18; Cervical Intraepithelial Neoplasia; Human Papillomavirus 16; Uterine Cervical Neoplasms
Keywords: Human Papillomavirus; Cervical Cancer; Screening
MeSH Terms: conditions — Uterine Cervical Dysplasia; Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Women referred to colposcopy clinic (Experimental): Triage tests for diagnosis of cervical pre-cancer amongHPV positive women
  Interventions: Device: OncoE6; Device: EVA System

INTERVENTIONS:
Device: OncoE6 — HPV oncoprotein assay
Device: EVA System — low-cost colposcope

SUMMARY:
Background:

* Cervical cancer is caused by persistent infection of the lining of the cervix with some kinds of human papillomaviruses (HPV). These HPV infections are distantly related to the viruses that cause warts on the skin. Like common wart viruses, most women who have cervical infections with HPV resolve the infections within 2 years without any need for treatment. Cervical infections that do not go away may cause disease that can turn into cancer after many years.
* Only one study has been done in Nigeria to learn how many women have HPV infection. The results of the study differed from most other studies in the world because older women were much more likely to be infected. This study with learn whether the results found in the previous study are true in Irun also, the site of the current study.

Objectives:

* To examine the age distribution of HPV infection and relationship to cancer of the cervix among Nigerian women.
* To understand how different screening methods, including HPV testing, could best reduce the risk of cervical cancer in Nigerian women.

Eligibility:

- Women residing in Irun, Nigeria, who are 15 years of age or older.

Design:

* Participants complete a brief questionnaire related to demographics, household and living conditions and a longer survey with questions related to reproductive history, family history, illnesses, stressful life events and sexual history (U. of Michigan collaboration).
* Participants have a cervical examination, HPV test, Pap test and blood test.
* Women whose tests show they are infected with HPV or have cervical disease will do the following:
* see a doctor and have cervical biopsies of all white abnormal areas (removal of a small tissue sample from the cervix)
* have photographs of the cervix taken
* have a cervical scraping for a new kind of HPV test.
* Some women with normal test results are also asked to see a doctor to check the validity of the testing
* Women with cervical disease receive treatment by a specialist and remain in the program until treatment is successfully completed or a final diagnosis is reached.
* Participants may be contacted for followup up to 5 years after the final diagnosis is made.

DETAILED DESCRIPTION:
BACKGROUND: Cervical cancer, caused by persistent infection with approximately 15-20 genotypes of carcinogenic human papillomavirus (HPV) infection, is the second leading cause of female cancer. Cytology (Pap smears) and the new HPV vaccines are not widely available in poor regions. Immediate treatment of HPV-infected older women by cryotherapy might have greater impact.

Although the same HPV types cause cervical cancer everywhere, and the same stages (infection, persistence vs. clearance, progression to precancer, and invasion) typify cervical carcinogenesis, the patterns of age-specific prevalence of HPV vary widely. These patterns are important for secondary prevention strategies relying on HPV DNA testing.

In many regions, including the US, HPV infections appear as classical sexually-transmitted agents, with peak cervical DNA prevalence at young ages (approximately 20) and low prevalence at older ages. However, in Nigeria, HPV prevalence is high (greater than or equal to 15%) at all ages according to the one study performed in urban Ibadan by Franceschi s group at IARC (n=932 women). This pattern is very uncommon. High prevalence at all ages would preclude use of HPV testing in low-cost strategies, due to poor positive predictive value. One possibly relevant element is the marital structure in Nigeria; a man often has multiple wives.

OBJECTIVES: The major objectives are: 1) To estimate age-specific HPV prevalences in Irun, Nigeria; 2) To investigate epidemiologic risk factors for HPV and cervical intraepithelial neoplasia in this population; 3) To examine the performance of screening options; 4) To assess the correlation of HPV among co-wives, comparing households with multiple wives with those with single wives; and 5) To validate the performance of rapid HPV, an inexpensive HPV test designed for public-sector use in settings like Irun.

ELIGIBILITY: All non-pregnant women aged 15+, without hysterectomy, will be eligible if they can provide written informed consent. Unmarried women less than 21 will be enrolled only with parental consent. Sexually active women will be examined and asked for cervical specimens; self-reported virginal women will be asked for a 10-ml blood sample only.

DESIGN: This is a cross-sectional screening study of 1500 women in Irun, a Nigerian village. Unlike the IARC study, we will incorporate cytology, visual inspection, and colposcopic biopsy of women that test positive by any of the three screening tests. We will determine whether HPV infection at various ages is related to risk of cervical abnormalities. The analyses will include descriptive trend data, multivariable modeling of HPV determinants, and clinical epidemiologic analysis of relative screening test performance in detecting cervical neoplasia.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Females who are 15 years to 99 years of age

EXCLUSION CRITERIA:

* Previous hysterectomy
* Current pregnancy
* Inability to give informed consent

Ages: 30 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1466 (Actual)
Dates: Start 2009-07-06 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-11-10 (Actual)

PRIMARY OUTCOMES:
Sensitivity of triage methods | cross-sectional
  Cervical Histopathology

CONTACTS AND LOCATIONS:
Overall Officials: Mark H Schiffman, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Obafemi Awolowo University Teaching Hospital, Ile-Ife, Nigeria

REFERENCES:
- [Background] Clarke MA, Gage JC, Ajenifuja KO, Wentzensen NA, Adepiti AC, Wacholder S, Burk RD, Schiffman M. A population-based cross-sectional study of age-specific risk factors for high risk human papillomavirus prevalence in rural Nigeria. Infect Agent Cancer. 2011 Jul 29;6:12. doi: 10.1186/1750-9378-6-12. PMID 21801395
- [Background] Gage JC, Ajenifuja KO, Wentzensen NA, Adepiti AC, Eklund C, Reilly M, Hutchinson M, Wacholder S, Harford J, Soliman AS, Burk RD, Schiffman M. The age-specific prevalence of human papillomavirus and risk of cytologic abnormalities in rural Nigeria: implications for screen-and-treat strategies. Int J Cancer. 2012 May 1;130(9):2111-7. doi: 10.1002/ijc.26211. Epub 2011 Aug 5. PMID 21630264
- [Background] Gage JC, Ajenifuja KO, Wentzensen N, Adepiti AC, Stoler M, Eder PS, Bell L, Shrestha N, Eklund C, Reilly M, Hutchinson M, Wacholder S, Castle PE, Burk RD, Schiffman M. Effectiveness of a simple rapid human papillomavirus DNA test in rural Nigeria. Int J Cancer. 2012 Dec 15;131(12):2903-9. doi: 10.1002/ijc.27563. Epub 2012 Apr 27. PMID 22473652